CLINICAL TRIAL: NCT05403151
Title: Controls and Healthy Vasculature Initiative
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000829; 000829-H
Record Dates: First submitted 2022-06-02; First posted 2022-06-03 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01-21

CONDITIONS: Vascular And Immunologic Diseases; Healthy Volunteers
Keywords: Sample Collection; Vascular; Blood; Inflammation; Thrombosis; Natural History
MeSH Terms: conditions — Inflammation; Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Healthy Adults

SUMMARY:
Background:

Diseases involving blood, blood vessels, and immune systems are leading causes of death in the United States. Researchers studying these diseases need to compare blood samples from both healthy and sick individuals. Blood samples from healthy people are also used to establish what is normal when developing new tests for diseases and to make sure new testing equipment is working properly.

Objective:

This natural history study will collect blood samples from healthy people. The blood will be used for various kinds of research.

Eligibility:

Healthy adults aged 18 years or older. Pregnant or nursing women will be excluded.

Design:

Participants will have a telehealth visit or telephone call to review their medical history.

They will come to the NIH Clinical Center. They will have a needle inserted into a vein in their arm or hand. About 10 tablespoons of blood will be drawn through the needle.

Researchers may perform a complete blood count, a type of blood test that can help evaluate the participant s overall health. They may do a blood type test.

The blood samples will also be used for genetic studies.

Some blood samples may be stored for use in future research.

Participants may choose to return for repeat visits for up to 10 years. Review of their medical history may also be repeated at later visits. They will receive $50 per blood collection visit.

...

DETAILED DESCRIPTION:
Study Description:

This study will serve to provide tissue samples from individuals with healthy vasculature for mechanistic studies of vascular inflammation and thrombosis.

Objectives:

Primary Objective:

To collect samples from healthy volunteers to:

* Establish and validate technical assays and equipment (e.g. platelet aggregation, inflammasome activation, neutrophil extracellular trap formation, tissue factor activity, etc.)
* Establish normal physiologic mechanisms and parameters in samples from healthy volunteers (e.g. platelet function, circulating autoantibody titers, etc.)

Endpoints:

This protocol does not have an outcome measure, but rather will be conducted in accordance with Good Clinical Practices for human research solely for the purpose of obtaining blood samples to optimize assays, conduct mechanistic investigations, measure vascular biomarkers, and facilitate the study of vascular and immunologic diseases in patients enrolled in other studies.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Stated willingness to comply with all study procedures
* Aged 18 years and older
* Ability of subject to understand and the willingness to sign a written informed consent document
* Self-reported in good general health

EXCLUSION CRITERIA:

An individual who, by self-report, meets the following criteria will be excluded from participation in this study:

-Current pregnancy or lactation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2032-01-30 (Estimated); Study Completion 2032-01-30 (Estimated)

PRIMARY OUTCOMES:
To collect samples from healthy volunteers to establish and validate technical assays and normal physiologic mechanisms and parameters for on-going and future basic and translational research studies. | Up to 10 Years
  This protocol does not have an outcome measure, but will obtain blood samples to optimize assays, conduct mechanistic investigations, measure vascular biomarkers, and facilitate the study of vascular and immunologic diseases in patients enrolled in other studies.

CONTACTS AND LOCATIONS:
Overall Officials: Yogendra Kanthi, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000829-H.html